CLINICAL TRIAL: NCT06225063
Title: The Comparison of Pilates with Cognitive Functional Therapy in Adults with Chronic Neck Pain: a Randomized Controlled Trial
Brief Title: The Comparison of Pilates with Cognitive Functional Therapy in Adults with Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University Cyprus (Other)
Responsible Party: Principal Investigator, Evi Lazoura, Physiotherapist, MSc, PhD (cand.), European University Cyprus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ΕΕΒΚ/ΕΠ/2023/20
Record Dates: First submitted 2024-01-13; First posted 2024-01-25 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-05

CONDITIONS: Chronic Neck Pain
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pilates Group (Experimental): In the first session participants will received the 6 basic principles of the technique. All the other sessions will last 50 minutes and consist of warm-up, main program and cool-down exercises. The degree of difficulty of the exercises of the main part will progress every 2 weeks.
  Interventions: Other: Pilates
- Cognitive Functional Therapy (Experimental): In this group the participants will receive personalized treatment and therefore the sessions will be done individually for each one. All interventions will include a) a cognitive component, b) specific functional training and c) lifestylwe changes
  Interventions: Other: Cognitive Functional Therapy

INTERVENTIONS:
Other: Pilates — The application of pilates aims to correct real-time deviations observed in the body during movement, to maintain stability, to maintain stability, to gradually form proper sensorimotor ability and improve cervical dysfunction. Pilates is an important part but also a primary point in the stages of rehabilitation, since through it the execution of movement is encouraged earlier thus providing help for the later stages of rehabilitation. Pilates exercises concern movements at all levels of body movement and in various positions.
  Other Names: pilates exercises
  Arms: Pilates Group
Other: Cognitive Functional Therapy — Cognitive component: Educating patients about their perceptions of pain, explaining diagnosis and diagnostic findings, answering questions about their problem and symptoms, progressively challenge their customers in a non-judgmental way, education for multifactorial and biopsychosocial spectrum of pain, encouraging participants to movement and for active participation in daily activities, if receiving a self-management plan participation in activities with a degree of difficulty 2-3/10, tips for more effective sleep Specific functional training: Understanding pain modification through relaxation exercises, awareness and body control, modified body positions for better control of the cervical spine with parallel relaxation of the thoracic spine to participate in fearful or painful activities, engaging in movements of daily activities Lifestyle changes: Gradual increase in physical activity based on patient preferences, stress management and social interaction
  Other Names: CFT
  Arms: Cognitive Functional Therapy

SUMMARY:
The aim of this study is to compare the effectiveness of Pilates compared with Cognitive Functional Therapy in adults with chronic neck pain.

DETAILED DESCRIPTION:
Firstly, people being informed about the study and those who determine eligibility criteria they written informer consent. After this, the participants will be randomized by a single-blind assessor in a 1:1 ration to pilates exercises and cognitive functional therapy. The participants of both groups will receive therapy twice a week for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64
* Pain in neck area for more than 3 months
* Pain in NPRS more than 40/100
* Independently mobility (with or without aid), to be capable of participating in a rehabilitation program twice a week

Exclusion Criteria:

* Serious psychological pathology
* Recently surgery on shoulder or neck area (<6 months)
* Pain relieving procedures such as injection based therapy and day case procedures (e.g. rhizotomy) in the last 3 months
* Pregnancy
* Rheumatologic/inflammatory disease (e.g. rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, lupus, Scheuermann's disease)
* Progressive neurological disease (e.g. Multiple Sclerosis, Parkinson's disease, Motor Neuron Disease)
* Unstable Cardiac Conditions
* Red flags disorders (malignancy/cancer, acute traumas like fracture (<6 months ago) or infection, spinal cord compression/cauda equina)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale | baseline (after randomization), at 4th week (after 8th session), at 8th week (after 16th session), 3 months after randomization
  Measured pain intensity with 0 (no pain) and 100 (the worst pain ever).
Neck Disability Index | baseline (after randomization), at 4th week (after 8th session), at 8th week (after 16th session), 3 months after randomization
  This questionnaire informed us about the affection to have the neck pain in human ability to manage it in everyday life. Measured neck disability with 4 (absence of disability) and >35 (full disability).

SECONDARY OUTCOMES:
Fear Avoidance Beliefs Questionnaire | baseline (after randomization), at 4th week (after 8th session), at 8th week (after 16th session), 3 months after randomization
  This questionnaire informed us how a patient's fear avoidance beliefs about physical activity and work may affect and contribute to their cervical pain and resulting disability, with 96 (high levels of patient fear) and 0 (absence of patient fear).
Short Form 12 | baseline (after randomization), at 4th week (after 8th session), at 8th week (after 16th session), 3 months after randomization
  This questionnaire assessed the impact of health on an individual's everyday life, with 0-42 indicates the possible existence of clinical depression and <42 indicates good psychological as well as physical functioning.
EuroQol (EQ-5D) | baseline (after randomization), at 4th week (after 8th session), at 8th week (after 16th session), 3 months after randomization
  An EQ-5D health state is the state of responses to the 5 dimensions of EQ-5D as completed by a patient, with 0 (the worst imaginable health state) and 100 (the best imaginable health state)
Range of Motion | baseline (after randomization), at 4th week (after 8th session), at 8th week (after 16th session), 3 months after randomization
  Range of motion in all cervical movements (flexion, extension, side flexion, rotations)
Isometric Strength | baseline (after randomization), at 4th week (after 8th session), at 8th week (after 16th session), 3 months after randomization
  Strength in all cervical movements (flexion, extension, side flexion, rotations)

CONTACTS AND LOCATIONS:
Overall Officials: Evi Lazoura, PhD (cand), Study Director — European University Cyprus
Locations (1):
- Evi Lazoura, Nicosia, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No